CLINICAL TRIAL: NCT01108705
Title: A Randomized, Double-blind, Multi-center Phase III Study of Brivanib Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Asian Subjects With Advanced Hepatocellular Carcinoma (HCC) Who Have Failed or Are Intolerant to Sorafenib
Brief Title: Comparison of Brivanib and Best Supportive Care (BSC) With Placebo and BSC for Treatment of Liver Cancer in Asian Patients Who Have Failed Sorafenib Treatment
Acronym: BRISK-APS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA182-047
Record Dates: First submitted 2010-04-15; First posted 2010-04-22 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — brivanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivanib (Experimental)
  Interventions: Drug: Brivanib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 800 mg, once daily, until disease progression or toxicity
  Other Names: BMS-582664
  Arms: Brivanib
Drug: Placebo — Tablets, Oral, 0mg, once daily, until disease progression or toxicity
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether brivanib is an effective treatment for liver cancer in Asian patients who have failed or could not tolerate sorafenib therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of advanced hepatocellular carcinoma
* Asian ethnicity
* Patient has failed ≥14 days of sorafenib treatment
* Cirrhotic status of Child-Pugh Class A or B with a score of 7
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Life expectancy of at least 8 weeks
* Adequate hematologic, hepatic, and renal function

Key Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy
* Previous or concurrent cancer that is distinct in primary site
* History of active cardiac disease
* Thrombotic or embolic events within the past 6 months
* Inability to swallow tablets or untreated malabsorption syndrome
* History of HIV infection
* Prior use of systemic investigational agents for hepatocellular carcinoma (except sorafenib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Compare overall survival of subjects with advanced HCC who have progressed on/after or are intolerant to sorafenib and receive brivanib plus best supportive care (BSC) to those receiving placebo plus BSC | Every 6 weeks for an average of 6 months

SECONDARY OUTCOMES:
Compare time to progression (TTP) using modified RECIST for HCC | Every 6 weeks
Compare objective response rate (ORR) and disease control rate (DCR) using modified RECIST for HCC | Every 6 weeks
Assess duration of response, duration of disease control and time to response | Every 6 weeks
Assess serious and nonserious adverse events, laboratory evaluations, significant physical examination findings and ECG results | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- China (18):
  - Local Institution, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Hankou, Hubei
  - Local Institution, Wuhan, Hubei
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Xi'an
- Local Institution, Singapore, Singapore
- South Korea (2):
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Taiwan (3):
  - Local Institution, Kaohsiung County
  - Local Institution, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx